CLINICAL TRIAL: NCT05771454
Title: Frequency of Occult Breast Cancer After Prophylactic Mastectomy Among High-Penetrance Breast Cancer Gene Positives; Future Implications on Sentinel Lymph Node Biopsy in LMIC: A Single-center Cross-sectional Study
Brief Title: Frequency of Occult Breast Cancer After Prophylactic Mastectomy Among High-Penetrance Breast Cancer Gene Positives
Acronym: OBC-PM
Status: Completed | Type: Observational
Sponsor: Aga Khan University Hospital, Pakistan (Other)
Responsible Party: Principal Investigator, Mehwish Mooghal , MBBS, Dr, Aga Khan University Hospital, Pakistan
Other Study IDs: 2022-8048-23560
Record Dates: First submitted 2023-03-06; First posted 2023-03-16 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Genetic Predisposition; BRCA Mutation; Breast Cancer; Occult Cancer
MeSH Terms: conditions — Genetic Predisposition to Disease; Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prophylactic risk reducing mastectomy: Patients who underwent genetic testing and came out positive for BRCA and other genes of breast cancer; afterwards opted for prophylactic risk-reducing mastectomy.
  After mastectomy, the specimens will be assessed for the presence of occult breast cancers in removed specimens. Histopathology is set as gold standard for occult breast cancer confirmation.
  Interventions: Procedure: Histopathological confirmation

INTERVENTIONS:
Procedure: Histopathological confirmation — After mastectomy, each specimen will be assessed histopathologically for the presence or absence of invasive focus of breast cancer.

SUMMARY:
The role of Sentinel Lymph Node Biopsy(SLNB) among mutation-negative BC patients is well established; however, we are lacking data to assess the role of sentinel lymph node biopsy for patients who are undergoing surgery for prophylactic reasons without proven malignancy. Literature has reported a positive Occult Breast Cancer (OBC) rate of 0 to 11.3% among mastectomy specimens which are removed prophylactically. Majority of the time when the invasive focus is diagnosed in prophylactic mastectomy specimens they are found to be in-situ cases where axillary Staging using SLNB can be exempted; however, when the OBC is identified even in prophylactic mastectomy specimens, axilla should be addressed accordingly. Albeit SLNB has associated complications with it; postoperative pain, lymphedema, paresthesia and rare reaction to the injected dye. Therefore the question here arises regarding skipping SLNB among patients who are undergoing PRRMs without proven malignancy pre-operatively. However, before standardizing the practice in our population we need convincing evidence that the frequency of OBC is low among our patients. By identifying the true prevalence of OBC among our gene-positive HBC patients who are opting for PRRM, we would be able to skip SLNB; as not only it has psychological implications but also adds a financial burden on patients and families due to the addition of an extra procedure and hospital bills; as the financial and socioeconomic status of our population has already declined over last few years due to the economic crises faced worldwide, specifically after-affects are seen in Lower Middle-Income Country(LMIC) like Pakistan.

DETAILED DESCRIPTION:
Recent studies have shown the rising incidence of Hereditary Breast Cancer (HBC) among Pakistani females, with growing numbers of Prophylactic Risk Reducing Mastectomies (PRRM) being offered to diagnosed cases of HBCs across different centres in the country.1 HBCs are seen in 5 to 10% of cases with Breast Cancers(BC). The main identified genes which contribute to the development of BCs among HBC patients are BRCA1, BRCA2, CDH1, PALB2, PTEN, TP53, ATM, BARD1, CHEK2, NF1, RAD51C/D and STK11. Among these culprit genes, BRCA1 and BRCA2 contribute to most HBC cases.

The role of Sentinel Lymph Node Biopsy(SLNB) among mutation-negative BC patients is well established; however, we are lacking data to assess the role of sentinel lymph node biopsy for patients who are undergoing surgery for prophylactic reasons without proven malignancy. Literature has reported a positive Occult Breast Cancer (OBC) rate of 0 to 11.3% among mastectomy specimens which are removed prophylactically. Majority of the time when the invasive focus is diagnosed in prophylactic mastectomy specimens they are found to be in-situ cases where axillary Staging using SLNB can be exempted; however, when the OBC is identified even in prophylactic mastectomy specimens, axilla should be addressed accordingly. Albeit SLNB has associated complications with it; postoperative pain, lymphedema, paresthesia and rare reaction to the injected dye. Therefore the question here arises regarding skipping SLNB among patients who are undergoing PRRMs without proven malignancy pre-operatively. However, before standardizing the practice in our population we need convincing evidence that the frequency of OBC is low among our patients. By identifying the true prevalence of OBC among our gene-positive HBC patients who are opting for PRRM, we would be able to skip SLNB; as not only it has psychological implications but also adds a financial burden on patients and families due to the addition of an extra procedure and hospital bills; as the financial and socioeconomic status of our population has already declined over last few years due to the economic crises faced worldwide, specifically after-affects are seen in Lower Middle-Income Country(LMIC) like Pakistan.

Due to the inflated cost and added procedure of SLNB in PRRM cases, our primary aim of this study is to evaluate the frequency of OBC among patients who underwent PRRMs concerning their high penetrance BC gene positivity; with the goal that SLNB can be safely omitted for PRRMs or not. Our secondary goal is to correlate the radiological findings with final histopathological results among OBC-positive patients, also the histopathological pattern of HBC genes among our cohort.

ELIGIBILITY:
Inclusion Criteria:

* individuals with positive genetic test results for High-Penetrance Hereditary BC genes, and those who had PRRMs at our center

Exclusion Criteria:

* individuals who did not give consent and those who had already diagnosed bilateral BCs

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All individuals who came out as genetic test positive for high-risk breast cancer genes; carriers/breast cancer patients and who opted for prophylactic risk-reducing mastectomy.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Occult breast cancer frequency | cross-sectional study. 2 months required for data collection from hospital records.
  frequency of identification of occult breast cancers among our cohort when prophylactic risk reducing mastectomy is done in mutation carriers.

CONTACTS AND LOCATIONS:
Locations (1):
- Aga Khan University Hospital, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No
If the data is to be shared, it will be shared in the form of an excel sheet without any patient identification.

REFERENCES:
- [Background] Sun YS, Zhao Z, Yang ZN, Xu F, Lu HJ, Zhu ZY, Shi W, Jiang J, Yao PP, Zhu HP. Risk Factors and Preventions of Breast Cancer. Int J Biol Sci. 2017 Nov 1;13(11):1387-1397. doi: 10.7150/ijbs.21635. eCollection 2017. PMID 29209143
- [Background] Daly M. B†, Pal T, Al Hilli Z, et al. Genetic/Familial High-Risk Assessment: Breast, Ovarian, and Pancreatic. NCCN Clinical Practice Guidelines in Oncology. Version 1.2023, 09/07/22 © 2022, [cited 2022 Sep 28]. Available from: https://www.nccn.org/guidelines/guidelines-detail
- [Background] Wong SM, Ferroum A, Apostolova C, Alhassan B, Prakash I, Basik M, Boileau JF, Meterissian S, Aleynikova O, Wong N, Foulkes WD. Incidence of Occult Breast Cancer in Carriers of BRCA1/2 or Other High-Penetrance Pathogenic Variants Undergoing Prophylactic Mastectomy: When is Sentinel Lymph Node Biopsy Indicated? Ann Surg Oncol. 2022 Oct;29(11):6660-6668. doi: 10.1245/s10434-022-11916-3. Epub 2022 May 26. PMID 35616744
- [Result] Akbar F, Siddiqui Z, Waheed MT, Ehsan L, Ali SI, Wiquar H, Valimohammed AT, Khan S, Vohra L, Zeeshan S, Rashid Y, Moosajee M, Jabbar AA, Zahir MN, Zahid N, Soomro R, Ullah NN, Ahmad I, Haider G, Ansari U, Rizvi A, Mehboobali A, Sattar A, Kirmani S. Spectrum of germline pathogenic variants using a targeted next generation sequencing panel and genotype-phenotype correlations in patients with suspected hereditary breast cancer at an academic medical centre in Pakistan. Hered Cancer Clin Pract. 2022 Jun 16;20(1):24. doi: 10.1186/s13053-022-00232-2. PMID 35710434